CLINICAL TRIAL: NCT03887026
Title: Efficacy and Safety of Single Doses of Norketotifen in Adult Subjects With Allergen-Induced Allergic Rhinitis in an Allergen Challenge Chamber
Brief Title: Efficacy and Safety of Norketotifen in Adults With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emergo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NKT-201
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Allergic Rhinitis; Allergic Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — norketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NKT Low Dose (Experimental): NKT single dose - Low
  Interventions: Drug: Norketotifen
- NKT High Dose (Experimental): NKT single dose - High
  Interventions: Drug: Norketotifen
- Placebo (Placebo Comparator): Placebo single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norketotifen — Norketotifen oral capsule
  Arms: NKT High Dose; NKT Low Dose
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
This is a Phase 2a study to evaluate the efficacy and safety of Norketotifen (NKT) in subjects with allergic rhinitis.

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized, placebo-controlled, 3-way crossover study evaluating the efficacy and safety of NKT in adult subjects with allergen-induced allergic rhinitis in an allergen challenge chamber.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide informed consent and comply with the protocol procedures
* Males and females, age 18 to 45 years, inclusive
* Other than seasonal allergic rhinitis, participant is healthy as determined by pre-study medical history, physical examination and vital signs. Any chronic conditions that may interfere with the study outcomes or the subject's safety will be considered clinically significant and a reason for exclusion.
* History of seasonal allergic rhinitis to mountain cedar pollen for at least the past 2 consecutive seasons
* Positive mountain cedar pollen skin prick test at Screening or within 12 months prior to Screening (wheal diameter ≥5 mm larger than the negative control)
* For females, negative serum pregnancy test. Females of childbearing potential and males must agree to use required contraception as outlined in the protocol

Exclusion Criteria:

* Female subjects who are pregnant or lactating
* Any history of epilepsy, diabetes mellitus, blood pressure abnormalities or cardiac arrhythmias
* Presence of any uncontrolled medical or psychiatric illness
* Treatment for controlled concurrent medical conditions has not been stable in terms of either doses or medications for at least 30 days prior to the baseline visit or is anticipated to change during the study
* Current use of or expected use of any of the prohibited medications within the indicated withholding timeframes as outlined in the protocol
* History of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Any history of malignancy within the past 5 years, with the exception of non-melanoma skin cancer
* History of pulmonary disease and/or active asthma requiring daily drug therapy. Mild, intermittent asthma is permitted (managed with short acting beta-agonist less than 3 times per week). Isolated exercise-induced bronchospasm is also permitted
* Any infection or inflammatory condition within the 2 weeks prior to screening
* Positive human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV) antibody screen
* Any clinically significant abnormal laboratory or ECG test. Presence of thrombocytopenia at screening is exclusionary
* Evidence of illicit drug use or positive urine Class A drug, alcohol, or cotinine screen
* Regular use of tobacco or nicotine containing products, including vaping, within 1 year prior to Screening
* Received any investigational drug within 30 days prior to Screening
* Any prior exposure to norketotifen
* History of allergic reaction to ketotifen
* In the opinion of the investigator, subject would be unlikely to comply with required study visits, self-assessments, and interventions

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score (TNSS) from pre-dose to 6 hours post-dose | 6 hours
  Change in TNSS from pre-dose to 6 hours post-dose for NKT vs placebo. The TNSS is the sum of the scores of four nasal symptoms (runny nose, congestion, itching, and sneezing) each scored on a scale of 0 to 3 (0=absent; 1=mild; 2=moderate; 3=severe). The TNSS score ranges from 0 to 12.

SECONDARY OUTCOMES:
Change in Total Ocular Symptom Score (TOSS) from pre-dose to 6 hours post-dose | 6 hours
  Change in TOSS from pre-dose to 6 hours post-dose for NKT vs placebo. The TOSS is the sum of the scores of three ocular symptoms (itching, tearing, and redness) each scored on a scale of 0 to 3 (0=absent; 1=mild; 2=moderate; 3=severe). The TOSS score ranges from 0 to 9.
Change in Total Symptom Score (TSS) from pre-dose to 6 hours post-dose | 6 hours
  Change in TSS from pre-dose to 6 hours post-dose for NKT vs placebo. The TSS is the sum of the TNSS and TOSS (described above) and ranges from 0 to 21.
Area under the curve (AUC) of TNSS over 6 hours post-dose | 6 hours
  AUC of TNSS over 6 hours post-dose for NKT vs placebo
AUC of TOSS over 6 hours post-dose | 6 hours
  AUC of TOSS over 6 hours post-dose for NKT vs placebo
AUC of TSS over 6 hours post-dose | 6 hours
  AUC of TSS over 6 hours post-dose for NKT vs placebo
Change in individual nasal symptoms from pre-dose to 6 hours post-dose | 6 hours
  Change in individual nasal symptoms from pre-dose to 6 hours post-dose for NKT vs placebo
Change in individual ocular symptoms from pre-dose to 6 hours post-dose | 6 hours
  Change in individual ocular symptoms from pre-dose to 6 hours post-dose for NKT vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Hazar Awad Granko, RPh, PhD, Study Chair — Emergo Therapeutics, Inc.
Locations (1):
- Biogenics Research Chamber, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No